CLINICAL TRIAL: NCT07192211
Title: Exploratory Study of ADR-002K for Heart Failure Patients With Ischemic Heart Disease Who Undergo Coronary Artery Bypass Surgery
Brief Title: Exploratory Study of ADR-002K for Heart Failure Patients With Ischemic Heart Disease Who Undergo CABG
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rohto Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADR-002K-0223
Record Dates: First submitted 2025-08-28; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal stem cell (Experimental)
  Interventions: Biological: Mesenchymal stem cell
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Mesenchymal stem cell — ADR-002K administration
  Arms: Mesenchymal stem cell
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
ADR-002K is administered to heart failure patients with ischemic heart disease who undergo coronary artery bypass surgery (CABG) to investigate its efficacy and safety.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled Phase II study. ADR-002K (Adipose-derived mesenchymal stem cells) is administered to the surface of the heart in patients with ischemic heart disease who undergo CABG. The efficacy and safety of ADR-002K are evaluated until the last patient has completed the 2-year evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients clinically diagnosed with chronic heart failure due to ischemic heart disease who undergo CABG
2. Patients with an LVEF of less than 40% as determined by the cardiac ultrasound at the screening examination.
3. Others

Exclusion Criteria:

1. Patients who have a combination of cardiovascular disease such as severe organic valvular disease.
2. Patients who have developed acute coronary syndrome within 3 months prior to obtaining consent.
3. Others

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Time to the first occurrence of the cardiovascular events | 2 years

SECONDARY OUTCOMES:
Left Ventricular Ejection Fraction (LVEF) in Cardiac MRI scan and Echocardiography | 2years
  Changes of LVEF in 2years after ADR-002K administration
Late Gadolinium Enhancement (LGE) in Cardiac MRI scan | 2 years
  Changes of LGE in the 2years after ADR-002K administration
Left Ventricular Remodeling in Cardiac MRI scan & Echocardiography | 2 years
  Changes of Left Ventricular End-Systolic Volume Index, Left Ventricular End-Diastolic Volume Index, Left Ventricular End-Systolic Diameter, Left Ventricular End-Diastolic Diameter) in 2 years after ADR-002K administration
6-minute walk distance | 2 years
  Changes of 6-minute walk distance in 2 years after ADR-002K administration
New York Heart Association | 2 years
  Changes of New York Heart Association in 2 years after ADR-002K administration
The Kansas City Cardiomyopathy Questionnaire（KCCQ) | 2 years
  Changes of KCCQ scores in 2 years after ADR-002K administration
Minesota Living With Heart Failure Questinanaire（MLHFQ） | 2 years
  Changes of MLHFQ scores in 2 years after ADR-002K administration
N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) | 2 years
  Changes of N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) in 2 years after ADR-002K administration
Adverse Events | 2 years
  Number and rate of adverse events related to this product

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Miyagawa, profesor, Principal Investigator — Osaka University

IPD SHARING:
Plan to Share IPD: No